CLINICAL TRIAL: NCT02535273
Title: The Effect of Dexmedetomidine Subsidiary Analgesia and Sedation in Minimally Invasive Spine Surgery Under Local Anesthesia：A Randomized, Double Blind Controlled Trial
Brief Title: The Effect of Dexmedetomidine Analgesia and Sedation in Minimally Invasive Spine Surgery Under Local Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tangdu-dex-loc
Record Dates: First submitted 2015-08-20; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Spinal Diseases; Local Anesthesia
Keywords: dexmedetomidine; prone position; spine surgery; Minimally invasive; local anesthesia
MeSH Terms: conditions — Spinal Diseases | interventions — Dexmedetomidine; Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low-dose Dexmedetomidine (Experimental): load dosage：Intravenous injection dexmedetomidine 1 µg/kg，completed within 10 minutes.
  Local anesthesia: lidocaine maintenance dose：Intravenous infusion of dexmedetomidine 0.3 μg/kg/min until the end of surgery
  Interventions: Drug: Dexmedetomidine; Drug: Lidocaine; Drug: Low-dose Dexmedetomidine
- Moderate-dose Dexmedetomidine (Experimental): load dosage：Intravenous injection dexmedetomidine 1 µg/kg，completed within 10 minutes.
  Local anesthesia: lidocaine maintenance dose：Intravenous infusion of dexmedetomidine 0.5 μg/kg/min until the end of surgery
  Interventions: Drug: Dexmedetomidine; Drug: Lidocaine; Drug: Moderate-dose Dexmedetomidine
- High-dose Dexmedetomidine (Experimental): load dosage：Intravenous injection dexmedetomidine 1 µg/kg，completed within 10 minutes.
  Local anesthesia: lidocaine maintenance dose：Intravenous infusion of dexmedetomidine 0.7 μg/kg/min until the end of surgery
  Interventions: Drug: Dexmedetomidine; Drug: Lidocaine; Drug: High-dose Dexmedetomidine
- normal saline Control group (Placebo Comparator): Intravenous injection normal saline equal quantity，completed within 10 minutes. Local anesthesia: lidocaine Intravenous infusion of normal saline 0.125 μg/kg/min until the end of surgery
  Interventions: Drug: Lidocaine; Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — load dosage：Intravenous injection dexmedetomidine 1 µg/kg，completed within 10 minutes.
  Other Names: Yisi
  Arms: High-dose Dexmedetomidine; Low-dose Dexmedetomidine; Moderate-dose Dexmedetomidine
Drug: Lidocaine — local anesthesia：0.67% lidocaine local anesthesia layer by layer to the periosteum at the puncture site，Establish puncture channel, injection 5ml 0.67% lidocaine into the vertebral body through the catheter, and observe 5-10min before operation
  Other Names: Lidocaine Hydrochloride Injection
Drug: Low-dose Dexmedetomidine — maintenance dose：Intravenous infusion of dexmedetomidine 0.3 μg/kg/min until the end of surgery
  Other Names: Yisi
  Arms: Low-dose Dexmedetomidine
Drug: Moderate-dose Dexmedetomidine — maintenance dose：Intravenous infusion of dexmedetomidine 0.5 μg/kg/min until the end of surgery
  Other Names: Yisi
  Arms: Moderate-dose Dexmedetomidine
Drug: High-dose Dexmedetomidine — maintenance dose：Intravenous infusion of dexmedetomidine 0.7 μg/kg/min until the end of surgery
  Other Names: Yisi
  Arms: High-dose Dexmedetomidine
Drug: normal saline — Intravenous injection normal saline equal quantity，completed within 10 minutes. Intravenous infusion of normal saline 0.125 μg/kg/min until the end of surgery
  Other Names: Sodium Chloride Physiological Solution
  Arms: normal saline Control group

SUMMARY:
Evaluate safety and efficacy of dexmedetomidine in minimally invasive spine surgery under local anesthesia sedation.Explore the appropriate concentration of dexmedetomidine, whether or not can reduce the amount of local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent；
* American Society of Anesthesiologists (ASA)classification:class I~II;Elective minimally invasive spine surgery；
* Age ≥18 years old, weighing 45 ~ 80 Kg, height 151 ~ 185 cm;
* hypertension within Ⅱ grade, or controlled with drugs within Ⅱ level；
* Diabetes fasting in 8.3mol/L or less

Exclusion Criteria:

* DEX allergy;
* Change anesthesia preoperative or intraoperative ;
* metabolic disorders, anemia has not been corrected;
* recent patients receiving sedatives and antidepressants;
* degenerative diseases of the central nervous elderly persons;
* serious central nervous system diseases (acute stroke, uncontrolled epilepsy, severe dementia);
* hypovolemia; 8) unstable angina or acute myocardial infarction;
* left ventricular ejection fraction less than 30%, heart rate lower than 45bpm;
* II-III degree heart block;
* acute hepatitis or severe liver disease (liver function C level);
* patients with renal insufficiency randomly assigned to receive treatment, but If patients need dialysis test is excluded or interruption ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Ramsay sedation score | From 1min before dexmedetomidine infusion to 2h after surgery，up to 4 hours
  Evaluation time point：1min before dexmedetomidine infusion；1min before local anesthesia；lidocaine infiltrate layer by layer to the periosteum，assessed up to 2min；Intraoperative most painful moments，assessed up to 5min；1min before returning to the ward；2h after surgery.Intraoperative most painful moments：nucleus pulpous probe or Balloon Dilatation.
visual analogue scale | From 1min before dexmedetomidine infusion to 2h after surgery，up to 4 hours
  Evaluation time point：1min before dexmedetomidine infusion；1min before local anesthesia；lidocaine infiltrate layer by layer to the periosteum，assessed up to 2min；Intraoperative most painful moments，assessed up to 5min；1min before returning to the ward；2h after surgery.Intraoperative most painful moments：nucleus pulpous probe or Balloon Dilatation.

SECONDARY OUTCOMES:
The total amount of lidocaine | 2h after surgery；
The patient and the surgeon satisfaction | 2h after surgery；
  four grades：Very satisfied; General satisfied; Not satisfied; Very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Sun Li, Principal Investigator — Air Force Military Medical University, China

REFERENCES:
- [Background] Nakamura Y, Yabuki S, Kikuchi S, Konno S. Minimally invasive surgery for osteoid osteoma of the cervical spine using microendoscopic discectomy system. Asian Spine J. 2013 Jun;7(2):143-7. doi: 10.4184/asj.2013.7.2.143. Epub 2013 May 22. PMID 23741555
- [Background] Smith N, Masters J, Jensen C, Khan A, Sprowson A. Systematic review of microendoscopic discectomy for lumbar disc herniation. Eur Spine J. 2013 Nov;22(11):2458-65. doi: 10.1007/s00586-013-2848-8. Epub 2013 Jun 23. PMID 23793558
- [Background] Yoshimoto M, Takebayashi T, Ida K, Tanimoto K, Yamashita T. Microendoscopic discectomy in athletes. J Orthop Sci. 2013 Nov;18(6):902-8. doi: 10.1007/s00776-013-0442-x. Epub 2013 Jul 20. PMID 23873279
- [Background] Gandhi SD, Anderson DG. Minimally invasive surgery for the lumbar spine. J Neurosurg Sci. 2012 Mar;56(1):27-34. PMID 22415380
- [Background] Arts MP. Reply to the letter to the editor of R. Q. Knight concerning "does minimally invasive lumbar disc surgery result in less muscle injury than conventional surgery? A randomized controlled trial" by M. Arts, R. Brand, et al. (2011) Eur Spine J 20(1):51-57. doi:10.1007/s00586-012-2491-9. Eur Spine J. 2013 Apr;22(4):899. doi: 10.1007/s00586-012-2643-y. Epub 2013 Jan 9. No abstract available. PMID 23299723